# Alcohol and Violence Prevention for College Students (ASAP)

NCT04089137

Informed Consent

March 4, 2021

# Georgia State University Information Statement

**Title:** +Change Norms Documentation

Principal Investigator: Amanda K. Gilmore, PhD

Co-Investigators: Lindsay Orchowski, PhD, Kelly Cue Davis, PhD, Debra Kaysen, PhD,

Ruschelle Leone, PhD, Dennis Reidy, PhD, and Katherine Masyn, PhD

Sponsor: National Institute on Alcoholism and Alcohol Abuse

# **Introduction and Key Information**

- You are invited to take part in a research study. It is up to you to decide if you would like to take part in the study.
- The purpose of this study is to understand alcohol use and sexual assault on your college campus.
- Your role in the study will last about 30 minutes during one session.
- You will be asked to do the following: complete a survey online.
- The risks of being in this study include: discomfort while completing the survey and loss of confidentiality.
- This study is not designed to benefit you. Overall, we hope to gain information about prevention programs for alcohol use and sexual assault for college students.
- If you do not wish to take part in this study, you do not have to.

## **Purpose**

The purpose of this study is to understand alcohol use and sexual assault at your college. You are being asked to participate in this project because the information you can provide to us will help us learn more about how we can improve our resource to prevent alcohol use and sexual assault at your college campus. You are invited to take part in this research study because you are a college student aged 18-25. A total of 6000 people will be invited to take part in this study, 3000 will be from Georgia State University and 3000 will be from Arizona State University.

## **Procedures**

If you decide to take part, you will complete a survey (~30 minutes) about alcohol use and sexual assault.

## **Future Research**

Researchers will remove information that may identify you and may use your data for future research. If we do this, we will not ask for any additional consent from you.

#### **Risks**

In this study, you will not have any more risks than you would in a normal day of life. No injury is expected from this study, but if you believe you have been harmed, contact the research team as soon as possible. Georgia State University and the research team have not set aside funds to compensate for any injury.

If you endorse suicidal ideation, you will be called by research staff to ensure your safety. If during the phone call, you are at acute risk for suicide then we will need to break confidentiality to ensure your safety.

#### **Benefits**

Version Date: March 4, 2021

This study is not designed to benefit you personally. Overall, we hope to gain information about alcohol use and sexual assault to inform prevention programs for college students.

# **Alternatives**

The alternative to taking part in this study is to not take part in the study.

# Compensation

If you were invited emailed from the list provided by the University Registrar, you will receive a \$15 gift card for participating in this study. If participating as part of the GSU SONA Subject Pool, you will receive .5 credit.

# Voluntary Participation and Withdrawal

You do not have to be in this study. If you decide to be in the study and change your mind, you have the right to drop out at any time. You may skip questions or stop participating at any time. This will not cause you to lose any benefits to which you are otherwise entitled.

# **Confidentiality**

We will keep your records private to the extent allowed by law. The following people and entities will have access to the information you provide:

- Study Investigators: : Lindsay Orchowski, PhD, Kelly Cue Davis, PhD, Debra Kaysen, PhD, Ruschelle Leone, PhD, Dennis Reidy, PhD, and Katherine Masyn, PhD
- GSU Institutional Review Board
- Office for Human Research Protection (OHRP)
- National Institute on Alcohol Abuse and Alcoholism

We will use a study number rather than your name on study records. The information you provide will be stored in a locked cabinet and/or on password- and firewall-protected computers. Data sent over the internet may not be secure. We will not collect IP addresses and all data collection is completed on websites with encryption to protect your identity. Your study number will be stored separately from the data to protect privacy. When we present or publish the results of this study, we will not use your name or other information that may identify you.

To help us protect your privacy, we have a Certificate of Confidentiality from the National Institutes of Health (NIH). With this Certificate, we can't be forced by a court order or subpoena to disclose information that could identify you in any civil, criminal, administrative, legislative or other proceeding.

There are circumstances where the Certificate doesn't protect against disclosure of your personally identifiable information:

- When the US government is inspecting or evaluating federally-funded studies
- When information must be disclosed to meet FDA requirements
- If you give someone written permission to receive research information or you voluntarily disclose your study information
- If the researcher reports that you threatened to harm yourself or others
- In cases of child abuse reported by the researcher
- If the investigator reports cases of contagious disease (such as HIV) to the state

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

### **Contact Information**

Contact Amanda K. Gilmore, PhD at 404-413-1416 or agilmore12@gsu.edu

- If you have questions about the study or your part in it
- If you have questions, concerns, or complaints about the study
- If you think you have been harmed by the study

The IRB at Georgia State University reviews all research that involves human participants. You can contact the IRB if you would like to speak to someone who is not involved directly with the study. You can contact the IRB for questions, concerns, problems, information, input, or questions about your rights as a research participant. Contact the IRB at 404-413-3500 or irb@gsu.edu.

You can print or save a copy of this form for your records.

If you agree to participate in this research, please click the continue button.